CLINICAL TRIAL: NCT03729362
Title: A Phase 3 Double-blind Randomized Study to Assess the Efficacy and Safety of Intravenous ATB200 Co-administered With Oral AT2221 in Adult Subjects With Late-onset Pompe Disease Compared With Alglucosidase Alfa/Placebo
Brief Title: A Study Comparing ATB200/AT2221 With Alglucosidase Alfa/Placebo in Adult Subjects With Late-onset Pompe Disease
Acronym: PROPEL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATB200-03
Record Dates: First submitted 2018-10-10; First posted 2018-11-02 (Actual); Results first posted 2023-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Pompe Disease (Late-onset)
Keywords: Pompe; rhGAA
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — miglustat; GAA protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cipaglucosidase Alfa/Miglustat (Experimental): Participants received cipaglucosidase alfa co-administered with miglustat every 2 weeks (Q2W).
  Interventions: Biological: Cipaglucosidase Alfa; Drug: Miglustat
- Alglucosidase Alfa/Placebo (Active Comparator): Participants received alglucosidase alfa co-administered with placebo Q2W.
  Interventions: Biological: Alglucosidase Alfa; Drug: Placebo

INTERVENTIONS:
Biological: Cipaglucosidase Alfa — Participants received an intravenous (IV) infusion dose over a 4-hour duration every 2 weeks (Q2W).
  Other Names: ATB200
  Arms: Cipaglucosidase Alfa/Miglustat
Drug: Miglustat — Participants received weight-based doses 1 hour prior to cipaglucosidase alfa infusion Q2W.
  Other Names: AT2221
  Arms: Cipaglucosidase Alfa/Miglustat
Biological: Alglucosidase Alfa — Participants received an IV infusion dose over a 4-hour duration Q2W.
  Other Names: Myozyme
  Arms: Alglucosidase Alfa/Placebo
Drug: Placebo — Miglustat matching placebo was administered orally 1 hour prior to alglucosidase alfa infusion Q2W.
  Arms: Alglucosidase Alfa/Placebo

SUMMARY:
This is a phase 3 double-blind randomized study to study the efficacy and safety of intravenous ATB200 Co-administered with oral AT2221 in adult subjects with Late Onset Pompe Disease compared with Alglucosidase Alfa/placebo.

DETAILED DESCRIPTION:
This is a double-blind, randomized, multicenter, international study of ATB200/AT2221 in adult subjects with late-onset Pompe disease (LOPD) who have received enzyme replacement therapy with alglucosidase alfa (ie, ERT-experienced) or who have never received ERT (ie, ERT naïve) compared with alglucosidase alfa/placebo.

The study will consist of a screening period up to 30 days, a 12-month treatment period, and a 30 day safety follow-up period. Subjects who complete this study will have the option to participate in an open label extension study to receive ATB200/AT2221 under a separate protocol.

Enzyme replacement therapy-experienced subjects will continue to take alglucosidase alfa during the screening period; treatment with alglucosidase alfa will then be replaced by study drug (ATB200/AT2221 or alglucosidase alfa/placebo) on the same schedule without interruption (ie, every 2 weeks).

Infusion visits will be scheduled every 2 weeks throughout the study; assessments (eg, clinical laboratory tests) for initial safety monitoring will be performed at these visits for the first 6 weeks of the study. Study visits that include efficacy, safety, and other assessments will be scheduled approximately every 3 months and may occur over 2 days, provided all study assessments and procedures (with the exception of pharmacokinetic [PK] sample collection) are performed before administration of study drug.

Efficacy assessments (ie, functional assessments) include evaluation of ambulatory function (6MWT), motor function tests (Gait, Stair, Gowers' maneuver, and Chair [GSGC] test and Timed Up and Go [TUG] test), muscle strength (manual muscle testing and quantitative muscle testing), and pulmonary function tests (forced vital capacity [FVC], slow vital capacity [SVC], maximal inspiratory pressure [MIP], maximal expiratory pressure [MEP], and sniff nasal inspiratory pressure [SNIP]). Patient reported outcomes (Rasch-built Pompe-specific Activity [R PAct] Scale, EuroQol 5 Dimensions 5 Levels Instrument [EQ-5D-5L], Patient-Reported Outcomes Measurement Information System [PROMIS®] instruments for physical function, fatigue, dyspnea, and upper extremity, and Subject's Global Impression of Change). The Physician's Global Impression of Change will also be performed.

Pharmacodynamic assessments include measurement of biomarkers of muscle injury (creatine kinase [CK]) and disease substrate (urinary hexose tetrasaccharide [Hex4]). Blood samples will be collected for determination of total GAA protein levels and AT2221 concentrations in plasma for a population PK analysis. Safety assessments include monitoring of adverse events (AEs), including infusion associated reactions (IARs), clinical laboratory tests (chemistry, hematology, and urinalysis), vital signs, physical examinations including weight, electrocardiograms (ECGs), and immunogenicity. Concomitant medications and nondrug therapies will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must provide signed informed consent prior to any study-related procedures being performed.
2. Male and female subjects are ≥ 18 years old and weigh ≥ 40 kg at screening.
3. Female subjects of childbearing potential and male subjects must agree to use medically accepted methods of contraception during the study and for 90 days after the last dose of study drug.
4. Subject must have a diagnosis of LOPD based on documentation of one of the following:

   1. deficiency of GAA enzyme
   2. GAA genotyping
5. Subject is classified as one of the following with respect to ERT status:

   1. ERT-experienced, defined as currently receiving standard of care ERT (alglucosidase alfa) at the recommended dose and regimen (ie, 20 mg/kg dose every 2 weeks) for ≥ 24 months
   2. ERT-naïve, defined as never having received investigational or commercially available ERT
6. Subject has a sitting FVC ≥ 30% of the predicted value for healthy adults (National Health and Nutrition Examination Survey III) at screening.
7. Subject performs two 6MWTs at screening that are valid, as determined by the clinical evaluator, and that meet all of the following criteria:

   1. both screening values of 6MWD are ≥ 75 meters
   2. both screening values of 6MWD are ≤ 90% of the predicted value for healthy adults
   3. the lower value of 6MWD is within 20% of the higher value of 6MWD

Exclusion Criteria

1. Subject has received any investigational therapy or pharmacological treatment for Pompe disease, other than alglucosidase alfa, within 30 days or 5 half-lives of the therapy or treatment, whichever is longer, before Day 1 or is anticipated to do so during the study.
2. Subject has received gene therapy for Pompe disease
3. Subject is taking any of the following prohibited medications within 30 days before Day 1:

   * miglitol (eg, Glyset)
   * miglustat (eg, Zavesca)
   * acarbose (eg, Precose or Glucobay)
   * voglibose (eg, Volix, Vocarb, or Volibo)

   Note: None of these medications have a half-life that, when multiplied by 5, is longer than 30 days.
4. Subject requires the use of invasive or noninvasive ventilation support for > 6 hours per day while awake.
5. Subject has a hypersensitivity to any of the excipients in ATB200, alglucosidase alfa, or AT2221.
6. Subject has a medical condition or any other extenuating circumstance that may, in the opinion of the investigator or medical monitor, pose an undue safety risk to the subject or may compromise his/her ability to comply with or adversely impact protocol requirements. This includes clinical depression (as diagnosed by a psychiatrist or other mental health professional) with uncontrolled or poorly controlled symptoms.
7. Subject, if female, is pregnant or breastfeeding at screening.
8. Subject, whether male or female, is planning to conceive a child during the study.
9. Subject does not have documentation of diagnosis of Pompe disease and refuses to undergo genetic testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-01-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (73):
- United States (25):
  - Neuromuscular Research Center, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California, Irvine, Irvine, California
  - UF Helath: University of Florida Clinical Research Center, Gainesville, Florida
  - University of South Florida Research Center, Tampa, Florida
  - Emory Clinic, Atlanta, Georgia
  - Indiana University Health Neuroscience Center, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Minnesota Clinical Research Unit, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Feinstein Institute for Medical Research, Manhasset, New York
  - NYU School of Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Neurology, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Health Science Center San Antonio, San Antonio, Texas
  - University of Utah, Center for Clinical and Translational Sciences, Salt Lake City, Utah
  - Lysosomal and Rare Disorders Research, Fairfax, Virginia
- Hospital Universitario Austral, Buenos Aires, Argentina
- Australia (4):
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre, Melbourne, Victoria
  - Westmead Hospital, Westmead
- Medizinische Universität Innsbruck, Innsbruck, Austria
- UZ Leuven, Leuven, Belgium
- University Clinical Centre of the Republic of Srpska, Banja Luka, Bosnia and Herzegovina
- UMHAT Alexandrovska, Sofia, Bulgaria
- Canada (2):
  - Heritage Medical Research Clinic, University of Calgary, Calgary, Alberta
  - McMaster University Medical Centre, Hamilton, Ontario
- Denmark (2):
  - Aarhus Universitets Hospital, Aarhus N
  - Rigshospitalet Copenhagen Neuromuscular Center, Copenhagen
- France (5):
  - Hôpital Neurologique Pierre Wertheimer, Bron
  - Hôpital Raymond Poincaré, Garches
  - Hôpital Salengro, Lille
  - Hôpital de la Timone, Marseille
  - Hôpital Pasteur, Nice
- Germany (4):
  - Friedrich-Baur Institut, Munich, Bavaria
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitätsklinikum Halle (Saale), Halle, Saxony-Anhalt
- Eginition Hospital, Athens, Attica, Greece
- Hungary (3):
  - Semmelweis University, Institute of Genomic Medicine and Rare Disease, Budapest
  - University of Pécs, Pécs
  - University of Szeged, Szeged
- Italy (2):
  - UOC di Neurologia e Malattie Neuromuscolari, Messina, NAP
  - UOC Genetica Medica, Napoli, NAP
- Japan (6):
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Fukuoka University Hospital, Fukuoka
  - Kagoshima University Hospital, Kagoshima
  - Izumi City General Hospital, Osaka
  - The Jikei University Hospital, Tokyo
  - National Center of Neurology and Psychiatry, Tokyo
- Erasmus MC, Rotterdam, Netherlands
- University of Auckland, Auckland, New Zealand
- Poland (2):
  - Szpital Uniwersytecki w Krakowie, Małogoskie
  - Centrum Medyczne, Rzeszów
- University Medical Centre Ljubljana, Ljubljana, Slovenia
- South Korea (2):
  - Pusan National University, Yangsan, Gyeongsangnam-do
  - Seoul National University Hospital, Seoul
- Hospital de la Santa Creu I Sant Pau, Barcelona, Spain
- Sahlgrenska University Hospital, Gothenburg, Sweden
- National Taiwan University Hospital, Taipei, Taiwan
- United Kingdom (4):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Cambridge University Hospitals, Cambridge
  - Royal Free Hospital NHS, London
  - Salford Royal NHS Foundation Trust, Salford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andersen H, Diaz-Manera J, Goker-Alpan O, Mozaffar T, Sitaraman Das S, Fox B, Amon F, O'Brien-Prince K, Goldman M, Holdbrook F, Jain V, Byrne BJ. Safety of home administration of cipaglucosidase alfa plus miglustat in late-onset Pompe disease: results from multiple clinical trials. Ther Adv Rare Dis. 2026 Jan 31;7:26330040261416943. doi: 10.1177/26330040261416943. eCollection 2026 Jan-Dec. PMID 41631150
- [Derived] Kushlaf H, Diaz-Manera J, Bratkovic D, Byrne BJ, Claeys KG, Clemens PR, Dimachkie MM, Kishnani PS, Laforet P, Roberts M, Schoser B, Toscano A, Castelli J, Holdbrook F, Sitaraman Das S, Goldman M, Mozaffar T; PROPEL Study Group. Switching Enzyme Replacement Therapy for Late-Onset Pompe Disease From Alglucosidase Alfa to Cipaglucosidase Alfa Plus Miglustat: Post Hoc Effect Size Analysis of PROPEL. Muscle Nerve. 2025 Aug;72(2):230-239. doi: 10.1002/mus.28420. Epub 2025 May 7. PMID 40342075
- [Derived] Kishnani PS, Byrne BJ, Claeys KG, Diaz-Manera J, Dimachkie MM, Kushlaf H, Mozaffar T, Roberts M, Schoser B, Hummel N, Kopiec A, Holdbrook F, Shohet S, Toscano A; PROPEL Study Group. Switching treatment to cipaglucosidase alfa plus miglustat positively affects patient-reported outcome measures in patients with late-onset Pompe disease. J Patient Rep Outcomes. 2024 Nov 13;8(1):132. doi: 10.1186/s41687-024-00805-w. PMID 39535661
- [Derived] MacCulloch A, Griffiths A, Johnson N, Shohet S. Health-Related Quality-of-Life Utility Values in Adults With Late-Onset Pompe Disease: Analyses of EQ-5D Data From the PROPEL Clinical Trial. J Health Econ Outcomes Res. 2024 Sep 18;11(2):80-85. doi: 10.36469/001c.121928. eCollection 2024. PMID 39318718
- [Derived] Kishnani PS, Shohet S, Raza S, Hummel N, Castelli JP, Sitaraman Das S, Jiang H, Kopiec A, Keyzor I, Hahn A. Validation of the Patient-Reported Outcomes Measurement Information System (PROMIS(R)) physical function questionnaire in late-onset Pompe disease using PROPEL phase 3 data. J Patient Rep Outcomes. 2024 Jan 31;8(1):13. doi: 10.1186/s41687-024-00686-z. PMID 38294575
- [Derived] Schoser B, Roberts M, Byrne BJ, Sitaraman S, Jiang H, Laforet P, Toscano A, Castelli J, Diaz-Manera J, Goldman M, van der Ploeg AT, Bratkovic D, Kuchipudi S, Mozaffar T, Kishnani PS; PROPEL Study Group. Safety and efficacy of cipaglucosidase alfa plus miglustat versus alglucosidase alfa plus placebo in late-onset Pompe disease (PROPEL): an international, randomised, double-blind, parallel-group, phase 3 trial. Lancet Neurol. 2021 Dec;20(12):1027-1037. doi: 10.1016/S1474-4422(21)00331-8. PMID 34800400

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 125 participants were randomized in the study at 62 clinical sites across 24 countries; 123 participants received at least 1 dose of study drug. Two participants randomized to the alglucosidase alfa/placebo group were never dosed because genotyping did not confirm the diagnosis of Pompe disease.
Groups:
- Cipaglucosidase Alfa/Miglustat: Cipaglucosidase alfa co-administered with miglustat every 2 weeks (Q2W).
- Alglucosidase Alfa/Placebo: Alglucosidase alfa co-administered with placebo Q2W.
Period: Overall Study
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Started | 85 | 40 (Two subjects randomized to this group never dosed because genotyping did not confirm diagnosis of Pompe disease.)
Received at Least 1 Dose of Study Drug | 85 | 38
Completed | 80 | 37
Not Completed | 5 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — COVID-19 Pandemic | 1 | 0
Not completed — Discontinued due to COVID-19 related pneumonia | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Genotyping did not confirm diagnosis of Pompe disease | 0 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of the study drug.
Groups:
- Cipaglucosidase Alfa/Miglustat: Cipaglucosidase alfa co-administered with miglustat Q2W.
- Total: Total of all reporting groups
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo | Total
Number analyzed (Participants) | 85 | 38 | 123
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 74 | 35 | 109
  >=65 years | 11 | 3 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (13.25) | 45.1 (13.30) | 46.8 (13.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 18 | 67
  Male | 36 | 20 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 1 | 1
  White | 74 | 30 | 104
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 52 in 6 Minute Walk Distance (6MWD)
Description: The efficacy of cipaglucosidase alfa/miglustat co-administration on ambulatory function was measured by the 6MWT. The 6MWD, measured in meters, is the distance walked on the 6MWT. A greater distance indicated greater endurance. An increase from baseline indicated improvement.
Time Frame: Baseline, Week 52
Population: Analysis was performed on Intent-to-treat (ITT)-observed (OBS) population. Number of participants analyzed are based on those who had 6MWD result at Week 52. In addition, 1 outlier subject in the alglucosidase alfa/placebo group was not included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: meter
Groups:
- Alglucosidase Alfa/Placebo: Alglucosidase alfa co-administered with placebo every 2 weeks (Q2W)
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 81 | 36
meter | 21.31 (11.56) | 7.10 (7.043)
Statistical Analysis 1: Comparison: Cipaglucosidase Alfa/Miglustat vs Alglucosidase Alfa/Placebo; The primary and key secondary endpoints were tested in hierarchical order as follows: The test for the primary endpoint was conducted first at the 1-sided 0.025 significance level, and if significant, the ordered key secondary endpoints were similarly tested. If at any point the null hypothesis for superiority failed to be rejected, then that comparison and any other comparison below it could not be claimed as successful and would be considered nominal; Test type: Superiority — Analysis used a mixed-effect model for repeated measures (MMRM). The model included terms for treatment, baseline 6MWD, age, height, weight (all as continuous covariates), enzyme replacement therapy (ERT) status (ERT-naïve versus ERT-experienced), gender, time, and treatment-by-time interaction. Time was used as a repeated measure, and an unstructured covariance approach was applied; p = 0.048, MMRM — 1-sided significance level of 0.025; LS Mean Difference = 14.21, 95% CI 2-sided [-2.6 to 31.02], Standard Error of Mean 8.481

2. Secondary Outcome: Change From Baseline to Week 52 in Sitting Forced Vital Capacity (FVC; % Predicted)
Description: The efficacy of cipaglucosidase alfa/miglustat co-administration on pulmonary function was measured by sitting FVC (% predicted). FVC is a standard pulmonary function test used to quantify respiratory muscle weakness.
Time Frame: Baseline, Week 52
Population: Analysis was performed on ITT-Last Observation Carried Forward (LOCF) population. In the cipaglucosidase alfa/miglustat group, 1 subject had no post-baseline values and was not included in the analysis. In the alglucosidase alfa/placebo group, the outlier subject was not included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: percentage of predicted FVC
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 84 | 37
percentage of predicted FVC | -1.04 (0.624) | -3.70 (0.953)
Statistical Analysis 1: Comparison: Cipaglucosidase Alfa/Miglustat vs Alglucosidase Alfa/Placebo; Change from baseline to Week 52 in sitting FVC was the first of 6 key secondary efficacy endpoints, which were analyzed according to a hierarchical order; Test type: Superiority — The analysis used an Analysis of Covariance (ANCOVA) model adjusted for the baseline value (as a continuous covariate) and ERT status (ERT-naïve versus ERT-experienced), as well as baseline age, gender, baseline height, and baseline weight; p = 0.012, ANCOVA — 1-sided significance level of 0.025; LS Mean Difference = 2.66, 95% CI 2-sided [0.37 to 4.95], Standard Error of Mean 1.156

3. Secondary Outcome: Change From Baseline to Week 52 in the Manual Muscle Test (MMT) Score for the Lower Extremities
Description: The total score for the MMT lower extremity strength included the following 8 body parts: right/left hip flexion, right/left hip abduction, right/left knee flexion and right/left knee extension. The MMT lower extremity score ranged from 0 to 40, with lower scores indicating weaker muscle strength. An increase from baseline indicated increased muscle strength.
Time Frame: Baseline, Week 52
Population: Analysis was performed on the ITT-LOCF population. In the cipaglucosidase alfa/miglustat group, 1 subject had neither baseline nor post-baseline values and 4 subjects had no post-baseline values; these subjects were not included in the analysis. In the alglucosidase alfa/placebo group, 3 subjects had neither baseline nor post-baseline values, and were not included in the analysis. In addition, the outlier subject was not included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 80 | 34
score on a scale | 1.64 (0.388) | 0.68 (0.603)
Statistical Analysis 1: Comparison: Cipaglucosidase Alfa/Miglustat vs Alglucosidase Alfa/Placebo; Change from baseline to Week 52 in the MMT score for the lower extremities was the second of 6 key secondary efficacy endpoints, which were analyzed according to a hierarchical order; Test type: Superiority — The analysis used an ANCOVA model adjusted for the baseline value (as a continuous covariate) and ERT status (ERT-naïve versus ERT-experienced), as well as baseline age, gender, baseline height, and baseline weight; p = 0.095, ANCOVA — 1-sided significance level of 0.025; LS Mean Difference = 0.96, 95% CI 2-sided [-0.48 to 2.4], Standard Error of Mean 0.727

4. Secondary Outcome: Change From Baseline to Week 26 in 6MWD
Description: The 6MWD, measured in meters, is the distance walked on the 6MWT.
Time Frame: Baseline, Week 26
Population: Analysis was performed on ITT-LOCF population. In the alglucosidase alfa/placebo group, the outlier subject was not included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: meter
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 85 | 37
meter | 16.45 (3.360) | 8.28 (5.168)
Statistical Analysis 1: Comparison: Cipaglucosidase Alfa/Miglustat vs Alglucosidase Alfa/Placebo; Change from baseline to Week 26 in 6MWD was the third of 6 key secondary efficacy endpoints, which were analyzed according to a hierarchical order; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.097, ANCOVA — 1-sided significance level of 0.025; LS Mean Difference = 8.17, 95% CI 2-sided [-4.24 to 20.57], Standard Error of Mean 6.261

5. Secondary Outcome: Change From Baseline to Week 52 in the Total Score for the Patient- Reported Outcomes Measurement Information System (PROMIS®) - Physical Function
Description: Physical Function Short Form 20a (v2.0) consisted of 20 questions. The first 14 questions were each scored on a scale from 1 to 5 as follows: 1 = unable to do; 2 = with much difficulty; 3 = with some difficulty; 4 = with a little difficulty; 5 = without any difficulty; the next 6 questions were each scored on a scale from 1 to 5 as follows: 1 = cannot do; 2 = quite a lot; 3 = somewhat; 4 = very little; 5 = not at all. The total score was calculated by summing up scores (1 to 5) across all items. Total scores range from 20 to 100. A higher score represented a better outcome.
Time Frame: Baseline, Week 52
Population: Analysis was performed on ITT-LOCF population. In the cipaglucosidase alfa/miglustat group, 1 subject had neither baseline nor post-baseline values, and was not included in the analysis. In the alglucosidase alfa/placebo group, the outlier subject was not included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 84 | 37
score on a scale | 1.98 (0.921) | 0.11 (1.406)
Statistical Analysis 1: Comparison: Cipaglucosidase Alfa/Miglustat vs Alglucosidase Alfa/Placebo; Change from baseline to Week 52 in the total score for the PROMIS® - Physical Function was the fourth of 6 key secondary efficacy endpoints, which were analyzed according to a hierarchical order; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.138, ANCOVA — 1-sided significance level of 0.025; LS Mean Difference = 1.87, 95% CI 2-sided [-1.51 to 5.25], Standard Error of Mean 1.706

6. Secondary Outcome: Change From Baseline to Week 52 in the Total Score for the PROMIS® - Fatigue
Description: Fatigue Short Form 8a consisted of 6 questions, each scored on a scale from 1 to 5 as follows: 1 = not at all; 2 = a little bit; 3 = somewhat; 4 = quite a bit; 5 = very much; and 2 questions, each scored on a scale from 1 to 5 as follows: 1 = never; 2 = rarely; 3 = sometimes; 4 = often; 5 = always. The total score was calculated by summing up scores (1 to 5) across all items. A lower score represented lower fatigue symptoms.
Time Frame: Baseline, Week 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 85 | 37
score on a scale | -1.90 (0.585) | -1.94 (0.901)
Statistical Analysis 1: Comparison: Cipaglucosidase Alfa/Miglustat vs Alglucosidase Alfa/Placebo; Change from baseline to Week 52 in the total score for the PROMIS® - Fatigue was the fifth of 6 key secondary efficacy endpoints, which were analyzed according to a hierarchical order; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.515, ANCOVA — 1-sided significance level of 0.025; LS Mean Difference = 0.04, 95% CI 2-sided [-2.12 to 2.2], Standard Error of Mean 1.092

7. Secondary Outcome: Change From Baseline to Week 52 in the Total Score for the Gait, Stairs, Gowers' Maneuver, and Chair (GSGC)
Description: The GSGC consisted of a 10-meter walk for evaluation of gait, a 4-stair climb, Gowers' maneuver, and arising from a chair. Results of the GSGC included the time required to complete the individual tests, individual scores for each of the tests (1 to 7 points for each of gait, 4-stair climb, and Gowers' maneuver, and 1 to 6 points for arising from a chair), and a total score. GSGC total score was the sum of the component scores from the 4 functional tests. The total score ranged from a minimum of 4 points (normal performance) to a maximum of 27 points (worst performance).
Time Frame: Baseline, Week 52
Population: Analysis was performed on ITT-LOCF population. In the cipaglucosidase alfa/miglustat group, 11 subjects had neither baseline nor post-baseline values, and 2 had no post-baseline values; these subjects were not included in the analysis. In the alglucosidase alfa/placebo group, 5 subjects had neither baseline nor post-baseline values, and 2 had no post-baseline values; these subjects were not included in the analysis. In addition, the outlier subject was not included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 72 | 30
score on a scale | -0.567 (0.280) | 0.847 (0.440)
Statistical Analysis 1: Comparison: Cipaglucosidase Alfa/Miglustat vs Alglucosidase Alfa/Placebo; Change from baseline to Week 52 in the total score for the GSGC was the sixth of 6 key secondary efficacy endpoints, which were analyzed according to a hierarchical order; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.004, ANCOVA — 1-sided significance level of 0.025; LS Mean Difference = -1.414, 95% CI 2-sided [-2.463 to -0.364], Standard Error of Mean 0.528

8. Secondary Outcome: Change From Baseline to Week 52 in Rasch-Built Pompe-Specific Activity (R-PAct) Total Score
Description: The R-PAct scale was an 18-item questionnaire to measure limitations in activities and restriction in social participation. Possible responses to questions were as follows: unable to perform, able to perform, but with difficulty, and able to perform without difficulty. The total score was calculated by summing up the observed scores across the 18 items and it ranged from 0 to 36, with higher values representing lower level of disease impact on the muscles.
Time Frame: Baseline, Week 52
Population: Analysis was performed on ITT-LOCF population. In the cipaglucosidase alfa/miglustat group, 16 subjects had neither baseline nor post-baseline values, and were not included in the analysis. In the alglucosidase alfa/placebo group, 4 subjects had neither baseline nor post-baseline values, and were not included in the analysis. In addition, the outlier subject was not included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 69 | 33
score on a scale | 0.04 (0.387) | 0.51 (0.567)

9. Secondary Outcome: Change From Baseline to Week 52 in European Quality of Life-5 Dimensions 5 Response Levels (EQ-5D-5L) Based on the EuroQol Visual Analogue Scale (EQ VAS) Quantitative Score
Description: The EuroQol Visual Analogue Scale (EQ VAS) is a vertical visual analogue scale that records the respondent's own assessment of his or her overall health status at the time of completion. Scores range from 0 (the worst health you can imagine) to 100 (the best health you can imagine). Higher EQ VAS scores represent an improved sense of overall health while lower scores represent a worsening of overall health.
Time Frame: Baseline, Week 52
Population: Analysis was performed on ITT-LOCF population. In the cipaglucosidase alfa/miglustat group, 1 subject had neither baseline nor post-baseline values, and was not included in the analysis. In the alglucosidase alfa/placebo group, 1 subject had neither baseline nor post-baseline values, and was not included in the analysis. In addition, the outlier subject was not included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 84 | 36
score on a scale | 0.03 (1.542) | 3.61 (2.400)

10. Secondary Outcome: Change From Baseline to Week 52 in Sitting Slow Vital Capacity (SVC) % Predicted
Description: SVC is a standard pulmonary function test used to quantify respiratory muscle weakness.
Time Frame: Baseline, Week 52
Population: Analysis was performed on ITT-LOCF population. In the cipaglucosidase alfa/miglustat group, 2 subjects had no post-baseline values and were not included in the analysis. In the alglucosidase alfa/placebo group, 1 subject had no baseline value, 1 subject had no post-baseline values, and they were not included in the analysis. In addition, the outlier subject was not included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: percentage of predicted SVC
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 83 | 35
percentage of predicted SVC | -2.527 (0.977) | -5.368 (1.527)

11. Secondary Outcome: Change From Baseline to Week 52 in Maximal Inspiratory Pressure (MIP) % Predicted
Description: The percent predicted values of MIP were calculated as: % predicted = (actual result / predicted result)* 100, where the predicted results were obtained using the reference equations from Uldry and Fitting (1995).
Time Frame: Baseline, Week 52
Population: Analysis was performed on ITT-LOCF population. In the cipaglucosidase alfa/miglustat group, 1 subject had no post-baseline value and was not included in the analysis. In the alglucosidase alfa/placebo group, the outlier subject was not included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: percentage of predicted MIP
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 84 | 37
percentage of predicted MIP | 1.89 (2.079) | -2.31 (3.178)

12. Secondary Outcome: Change From Baseline to Week 52 in Maximal Expiratory Pressure (MEP) % Predicted
Description: The percent predicted values of MEP were calculated as: % predicted = (actual result / predicted result)
  * 100, where the predicted results were obtained using the reference equations from Uldry and Fitting (1995).
Time Frame: Baseline, Week 52
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: percentage of predicted MEP
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 84 | 37
percentage of predicted MEP | 0.51 (1.996) | -1.35 (3.052)

13. Secondary Outcome: Change From Baseline to Week 52 in Sniff Nasal Inspiratory Pressure (SNIP) % Predicted
Description: The percent predicted values of SNIP were calculated as: % predicted = (actual result / predicted result) * 100, where the predicted results were obtained using the reference equations from Evans and Whitelaw (2009).
Time Frame: Baseline, Week 52
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: percentage of predicted SNIP
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 84 | 37
percentage of predicted SNIP | 1.40 (1.918) | 4.53 (2.929)

14. Secondary Outcome: Change From Baseline to Week 52 in % Predicted 6MWD
Description: The % predicted 6MWD = (actual 6MWD / predicted 6MWD) * 100. The predicted values were calculated using Enright And Sherrill 1998 Reference Equations.
Time Frame: Baseline, Week 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percentage of predicted 6MWD
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 85 | 37
percentage of predicted 6MWD | 4.039 (0.716) | 1.655 (1.102)

15. Secondary Outcome: Change From Baseline to Week 52 in the Quantitative Muscle Test (QMT) Values
Description: QMT was measured using the hand-held dynamometer. Larger values (in kg) indicated greater muscle strength.
Time Frame: Baseline, Week 52
Population: Analyses were performed on ITT-LOCF population. Number of participants analyzed for each of the QMT parameters displayed are based upon the number of participants who had both baseline and post-baseline values for each respective QMT parameter. In addition, the outlier subject in the alglucosidase alfa/placebo group was not included in the analyses.
Measure: Least Squares Mean (Standard Error); unit: kilogram
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 85 | 37
kilogram
  QMT Value for the Upper Extremities: number analyzed (Participants) | 83 | 37
  QMT Value for the Upper Extremities | 1.839 (2.098) | -0.553 (3.195)
  QMT Value for the Lower Extremities: number analyzed (Participants) | 81 | 36
  QMT Value for the Lower Extremities | 6.496 (3.185) | 5.265 (4.854)
  QMT Total Value: number analyzed (Participants) | 81 | 36
  QMT Total Value | 8.195 (5.079) | 5.198 (7.746)
  QMT Value for the Proximal Muscle Group: number analyzed (Participants) | 82 | 36
  QMT Value for the Proximal Muscle Group | 3.401 (2.920) | 0.945 (4.477)

16. Secondary Outcome: Change From Baseline to Week 52 in Other MMT Scores
Description: Each manual muscle test was evaluated on a scoring scale from 0 to 5, as follows: 0 = no muscle movement; 1 = visible muscle movement, but no movement at the joint; 2 = movement at the joint, but not against gravity; 3 = movement against gravity, but not against added resistance; 4 = movement against resistance, but less than normal; 5 = normal strength. Upper extremity score was the sum of scores for right/left shoulder abduction, right/left shoulder adduction, right/left elbow extension, and right/left elbow flexion, with the total score ranging from 0 to 40.
  Proximal muscle group score, the sum of scores for right/left hip flexion, right/left hip abduction, right/left shoulder abduction, and right/left shoulder adduction, with the total score ranging from 0 to 40. MMT total score was the sum of the lower and upper extremity scores and ranged from 0 to 80. Lower scores indicated lower overall muscle strength. An increase from baseline indicated improvement in muscle strength.
Time Frame: Baseline, Week 52
Population: Analyses were performed on ITT-LOCF population. Number of participants analyzed for each of the MMT parameters displayed are based upon the number of participants who had both baseline and post-baseline values for each respective MMT parameter. In addition, the outlier subject in the alglucosidase alfa/placebo group was not included in the analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 85 | 37
score on a scale
  MMT Upper Extremity Score: number analyzed (Participants) | 83 | 37
  MMT Upper Extremity Score | 1.54 (0.323) | 0.60 (0.491)
  MMT Total Score: number analyzed (Participants) | 80 | 34
  MMT Total Score | 3.24 (0.622) | 1.02 (0.966)
  MMT Proximal Muscle Group Score: number analyzed (Participants) | 81 | 36
  MMT Proximal Muscle Group Score | 1.82 (0.393) | 0.70 (0.599)

17. Secondary Outcome: Change From Baseline to Week 52 in Maximum Vital Capacity (Maximum VC) % Predicted
Description: Maximum VC is the greater of the two VC values (FVC or SVC).
Time Frame: Baseline, Week 52
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: percentage of predicted maximum VC
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 84 | 37
percentage of predicted maximum VC | -1.286 (0.613) | -3.695 (0.936)

18. Secondary Outcome: Change From Baseline to Week 52 in PROMIS-Dyspnea and Upper Extremities Total Scores
Description: The Upper Extremities Short Form 7a consisted of 7 items each scored on a decreasing scale from 1 to 5 as follows: 1 = unable to do; 2 = with much difficulty; 3 = with some difficulty; 4 = with a little difficulty; 5 = without any difficulty.
  Dyspnea Severity Short Form 10a consisted of 10 items each scored on a scale from 0 to 3 as follows: 0
  = no shortness of breath; 1 = mildly short of breath; 2 = moderately short of breath; 3 = severely short of breath.
  A total score was generated for each instrument by adding up each item. Total scores for upper extremities range from 7 to 35. Total scores for dyspnea range from 0 to 30. A higher score for upper extremities represented improvement in symptoms. A lower score for dyspnea severity represented improvement in symptoms.
Time Frame: Baseline, Week 52
Population: Analyses were performed on ITT-LOCF population. Number of participants analyzed for each of the PROMIS total scores displayed are based upon the number of participants who had both baseline and post-baseline values for each respective PROMIS total score (PROMIS-Dyspnea and Upper Extremities Total Scores). In addition, the outlier subject in the alglucosidase alfa/placebo group was not included in the analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 85 | 37
score on a scale
  PROMIS-Dyspnea Total Score: number analyzed (Participants) | 82 | 36
  PROMIS-Dyspnea Total Score | -0.41 (0.426) | -1.50 (0.652)
  PROMIS-Upper Extremities Total Score: number analyzed (Participants) | 84 | 37
  PROMIS-Upper Extremities Total Score | 0.97 (0.545) | 0.87 (0.833)

19. Secondary Outcome: Change From Baseline in the Time to Complete Individual GSGC Component Tests and Timed Up and Go (TUG) Test at Week 52
Description: Motor function test assessed the time to complete individual GSGC component tests (10-meter walk, 4- stair climb, Gowers' maneuver, and arise from a chair) and the TUG test. The TUG test assessed the time a subject needed to rise from a chair, walk 3 meters, turn around, walk back to the chair, and sit down.
Time Frame: Baseline, Week 52
Population: Analyses were performed on ITT-LOCF population. Number of participants analyzed for each of the GSGC components and the TUG test displayed are based upon the number of participants who had both baseline and post-baseline values for each respective GSGC component and the TUG test. In addition, the outlier subject in the alglucosidase alfa/placebo group was not included in the analyses.
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 85 | 37
seconds
  Time to complete the 10-meter walk: number analyzed (Participants) | 80 | 35
  Time to complete the 10-meter walk | -0.60 (0.631) | 2.06 (0.967)
  Time to complete the 4-stair climb: number analyzed (Participants) | 78 | 34
  Time to complete the 4-stair climb | -6.75 (0.851) | -3.61 (1.308)
  Time to complete the Gowers' maneuver: number analyzed (Participants) | 61 | 25
  Time to complete the Gowers' maneuver | -0.36 (0.799) | -1.95 (1.281)
  Time to arise from a chair: number analyzed (Participants) | 77 | 32
  Time to arise from a chair | -7.57 (0.409) | -6.75 (0.643)
  Time to complete the timed up and go test: number analyzed (Participants) | 75 | 31
  Time to complete the timed up and go test | -0.39 (0.768) | 0.09 (1.217)

20. Secondary Outcome: Physician's Global Impression of Change (PGIC) Overall Status at Week 52
Description: Physician's Global Impression of Change is based on a single item that is scored on a 7-point rating scale ranging from 1 "very much worse" to 7 "very much improved".
  A tertiary response variable (improving, declining, stable) was defined as follows: "Improving", which consisted of improved, moderately improved, and very much improved; "Declining", which consisted of worse, moderately worse, and very much worse; and "Stable", which equaled to no change.
Time Frame: Week 52
Population: Analysis was performed on ITT-OBS population. Number of participants analyzed are based on those who had PGIC data at Week 52. In addition, the outlier subject in the alglucosidase alfa/placebo group was not included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 80 | 36
Participants
  Improving | 31 | 10
  Stable | 38 | 16
  Declining | 11 | 10

21. Secondary Outcome: Subject's Global Impression of Change (SGIC) at Week 52
Description: The SGIC is designed to record the participants' impression of their functional status since starting study drug using a 7-point scale ranging from 1 "very much worse" to 7 "very much improved".
  A tertiary response variable (improving, declining, stable) was defined as follows: "Improving", which consisted of improved, moderately improved, and very much improved; "Declining", which consisted of worse, moderately worse, and very much worse; and "Stable", which equaled to no change.
Time Frame: Week 52
Population: Analysis was performed on ITT-OBS population. Number of participants analyzed are based on those who had SGIC data at Week 52. In addition, the outlier subject in the alglucosidase alfa/placebo group was not included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 81 | 36
Participants
  Improving | 36 | 13
  Stable | 33 | 12
  Declining | 12 | 11

22. Secondary Outcome: Number of Participants Improving on Both 6MWD and % Predicted FVC at Week 52
Description: A composite subject-level response of the 2 relevant clinical outcomes, 6MWD and FVC (% predicted), was assessed. Prespecified thresholds were used for assessment of improvement consistent with published minimal clinically important difference values for comparable instruments in similar disease.
Time Frame: Week 52
Population: Analysis was performed on ITT-LOCF population. In the cipaglucosidase alfa/miglustat group, 1 subject who had no post-baseline FVC value was counted as not improved and included in the analysis. In the alglucosidase alfa/placebo group, the outlier subject was not included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 85 | 37
Participants | 14 | 0

23. Secondary Outcome: Number of Participants With Treatment-Emergent Anti-Drug Antibodies (ADAs)
Description: Treatment-emergent ADAs were defined as participants who had seroconverted or boosted their preexisting ADA during the study period.
Time Frame: Baseline up to Week 52
Population: Analysis was performed on safety population which included subjects who had received at least 1 dose of study drug. Number analyzed equals participants evaluable at specified treatment.
Measure: Number; unit: participants
Groups:
- Cipaglucosidase Alfa/Miglustat: Participants who were exposed to at least 1 dose of cipaglucosidase alfa/miglustat.
- Alglucosidase Alfa/Placebo: Participants who were exposed to at least 1 dose of alglucosidase alfa/placebo.
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 85 | 38
participants
  ERT-experienced: Treatment-emergent ADAs: number analyzed (Participants) | 65 | 30
  ERT-experienced: Treatment-emergent ADAs | 31 | 5
  ERT-naïve: Treatment-emergent ADAs: number analyzed (Participants) | 20 | 8
  ERT-naïve: Treatment-emergent ADAs | 19 | 8

24. Secondary Outcome: Change From Baseline to Week 52 in Urinary Hexose Tetrasaccharide (Hex4) Level
Description: Levels of urinary Hex4, a biomarker of disease substrate, were measured. The assay specifically targets Hex4, the glucose tetrasaccharide (Glc4), which is a biomarker of glycogen storage.
Time Frame: Baseline, Week 52
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mmol/mol creatinine
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 84 | 37
mmol/mol creatinine | -1.88 (2.380) | 1.22 (4.432)

25. Secondary Outcome: Change From Baseline to Week 52 in Serum Creatine Kinase (CK) Level
Description: Change from baseline to Week 52 in serum CK level. CK levels were measured as part of the serum chemistry panel.
Time Frame: Baseline, Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 85 | 37
U/L | -130.5 (231.18) | 60.2 (159.49)

26. Secondary Outcome: Population Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of Cipaglucosidase Alfa and Alglucosidase Alfa in ERT-Experienced Participants Using Plasma Total GAA Protein Level by Signature Peptide Assay and Plasma Miglustat Concentration
Description: On Days 1 and 364 (Week 52), sparse blood samples were collected for PK analysis in ERT-experienced participants at 0, 1, 4, 6, 12, and 24 hours post-dose. Collection of the 12-hour sample was optional.
Time Frame: Days 1 and 364 (Week 52)
Population: Number analyzed equals participants evaluable at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Groups:
- Cipaglucosidase Alfa/Miglustat: Participants who were exposed to at least 1 dose of cipaglucosidase alfa/miglustat and had at least 1 PK assessment.
- Alglucosidase Alfa/Placebo: Participants who were exposed to at least 1 dose of alglucosidase alfa/placebo and had at least 1 PK assessment.
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 56 | 26
μg/mL
  Day 1 | 280 (18.5) | 289 (13.2)
  Day 364: number analyzed (Participants) | 44 | 21
  Day 364 | 293 (19.9) | 283 (17.6)

27. Secondary Outcome: Population PK: Area Under the Concentration-Time Curve (AUC) of Cipaglucosidase Alfa and Alglucosidase Alfa in ERT-Experienced Participants Using Plasma Total GAA Protein Level by Signature Peptide Assay and Plasma Miglustat Concentration
Description: as for outcome 26
Time Frame: Days 1 and 364 (Week 52)
Population: Number analyzed equals participants evaluable at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg·h/mL
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 56 | 26
μg·h/mL
  Day 1 | 1395 (21.5) | 1700 (17.6)
  Day 364: number analyzed (Participants) | 26 | 21
  Day 364 | 1476 (21.8) | 1688 (23.9)

28. Secondary Outcome: Population PK: Cmax of Cipaglucosidase Alfa and Alglucosidase Alfa in ERT-Naïve Participants
Description: On Days 1 and 364 (Week 52), sparse blood samples were collected for PK analysis in ERT-naïve participants at 0, 1, 4, 6, 12, and 24 hours post-dose. Collection of the 12-hour sample was optional.
Time Frame: Days 1 and 364 (Week 52)
Population: Number analyzed equals participants evaluable at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 18 | 7
μg/mL
  Day 1 | 273 (18.1) | 342 (31.0)
  Day 364: number analyzed (Participants) | 16 | 7
  Day 364 | 290 (17.4) | 359 (28.1)

29. Secondary Outcome: Population PK: AUC of Cipaglucosidase Alfa and Alglucosidase Alfa in ERT-Naïve Subjects
Description: as for outcome 28
Time Frame: Days 1 and 364 (Week 52)
Population: Number analyzed equals participants evaluable at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg·h/mL
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
Number analyzed (Participants) | 18 | 7
μg·h/mL
  Day 1 | 1343 (25.7) | 1859 (22.4)
  Day 364: number analyzed (Participants) | 16 | 7
  Day 364 | 1457 (19.2) | 1964 (26.8)

30. Secondary Outcome: Noncompartmental Analysis: Cmax of Plasma Total GAA Protein by Signature Peptide T09 in ERT-Naïve Subjects
Description: A noncompartmental analysis was performed on ERT-naïve subjects, who underwent serial PK sampling during the study. On Day 1, serial blood samples were collected for ERT-naïve participants just prior to initiation of cipaglucosidase alfa/alglucosidase alfa infusion (time 0) and at 1, 2, 3, 3.5, 4, 4.5, 6, 8, 10, and 24 hours after the start of cipaglucosidase alfa/alglucosidase alfa infusion for plasma total human acid α-glucosidase (GAA) protein signature peptide T09 and plasma miglustat determinations.
Time Frame: Day 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Groups:
- Cipaglucosidase Alfa: Participants who were exposed to at least 1 dose of cipaglucosidase alfa and had at least 1 PK assessment.
- Alglucosidase Alfa: Participants who were exposed to at least 1 dose of alglucosidase alfa and had at least 1 PK assessment.
- Miglustat: Participants who were exposed to at least 1 dose of miglustat and had at least 1 PK assessment.
Arm/Group | Cipaglucosidase Alfa | Alglucosidase Alfa | Miglustat
Number analyzed (Participants) | 12 | 4 | 12
μg/mL | 260 (18.4) | 364 (66.7) | 2768 (30.8)

31. Secondary Outcome: Noncompartmental Analysis: AUC From Time 0 (Predose) to the Time of Last Quantifiable Concentration of Plasma Total GAA Protein by Signature Peptide T09 in ERT-Naïve Subjects
Description: A noncompartmental analysis was performed on ERT-naïve subjects, who underwent serial PK sampling during the study. On Day 1, serial blood samples were collected for ERT-naïve participants just prior to initiation of cipaglucosidase alfa/alglucosidase alfa infusion (time 0) and at 1, 2, 3, 3.5, 4, 4.5, 6, 8, 10, and 24 hours after the start of cipaglucosidase alfa/alglucosidase alfa infusion for plasma total GAA protein signature peptide T09 and plasma miglustat determinations.
Time Frame: Day 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg·h/mL
Arm/Group | Cipaglucosidase Alfa | Alglucosidase Alfa | Miglustat
Number analyzed (Participants) | 12 | 4 | 12
μg·h/mL | 1264 (28.9) | 1656 (28.9) | 20588 (36.8)

32. Secondary Outcome: Comparison of Cmax of Cipaglucosidase Alfa in ERT-Experienced and ERT-Naïve Populations
Description: On Days 1 and 364 (Week 52), sparse blood samples were collected for PK analysis at 0, 1, 4, 6, 12, and 24 hours post-dose. Collection of the 12-hour sample was optional.
Time Frame: Days 1 and 364 (Week 52)
Population: Number analyzed based upon number of subjects with evaluable data for population PK analysis at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Groups:
- Cipaglucosidase Alfa (ERT-experienced): ERT-experienced participants who were exposed to at least 1 dose of cipaglucosidase alfa and had at least 1 PK assessment.
- Cipaglucosidase Alfa (ERT-naive): ERT-naive participants who were exposed to at least 1 dose of cipaglucosidase alfa and had at least 1 PK assessment.
Arm/Group | Cipaglucosidase Alfa (ERT-experienced) | Cipaglucosidase Alfa (ERT-naive)
Number analyzed (Participants) | 56 | 18
μg/mL
  Day 1 | 280 (18.5) | 273 (18.1)
  Day 364: number analyzed (Participants) | 44 | 16
  Day 364 | 296 (19.9) | 290 (17.4)

33. Secondary Outcome: Comparison of AUC of Cipaglucosidase Alfa in ERT- Experienced and ERT-Naïve Populations
Description: as for outcome 32
Time Frame: Days 1 and 364 (Week 52)
Population: Number analyzed based upon number of subjects with evaluable data for population PK analysis at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg·h/mL
Arm/Group | Cipaglucosidase Alfa (ERT-experienced) | Cipaglucosidase Alfa (ERT-naive)
Number analyzed (Participants) | 56 | 18
μg·h/mL
  Day 1 | 1395 (21.5) | 1343 (25.7)
  Day 364: number analyzed (Participants) | 44 | 16
  Day 364 | 1476 (21.8) | 1457 (19.2)

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) through Week 52 and follow-up (30 days after last dose).
Groups:
- Cipaglucosidase Alfa/Miglustat: All participants who received at least 1 dose of study drug (cipaglucosidase alfa/miglustat).
- Alglucosidase Alfa/Placebo: All participants who received at least 1 dose of study drug (alglucosidase alfa/placebo).
Arm/Group | Cipaglucosidase Alfa/Miglustat | Alglucosidase Alfa/Placebo
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/38
Serious Adverse Events (participants affected / at risk) | 8/85 | 1/38
Other Adverse Events (participants affected / at risk) | 69/85 | 32/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cipaglucosidase Alfa/Miglustat (N=85) | Alglucosidase Alfa/Placebo (N=38)
Aortic aneurysm (Vascular disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Ilium fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Removal of internal fixation (Surgical and medical procedures) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Anaphylactoid reaction (Immune system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Viral myositis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cipaglucosidase Alfa/Miglustat (N=85) | Alglucosidase Alfa/Placebo (N=38)
Hypertension (Vascular disorders) | 5 | 3
Contusion (Injury, poisoning and procedural complications) | 5 | 3
Fall (Injury, poisoning and procedural complications) | 25 | 15
Limb injury (Injury, poisoning and procedural complications) | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 2
Balance disorder (Nervous system disorders) | 1 | 2
Dizziness (Nervous system disorders) | 8 | 3
Headache (Nervous system disorders) | 20 | 9
Asthenia (General disorders) | 1 | 4
Fatigue (General disorders) | 8 | 5
Infusion site bruising (General disorders) | 1 | 2
Infusion site erythema (General disorders) | 0 | 2
Pain (General disorders) | 6 | 1
Pyrexia (General disorders) | 6 | 1
Panic attack (Psychiatric disorders) | 2 | 2
Abdominal distension (Gastrointestinal disorders) | 5 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 4 | 3
Constipation (Gastrointestinal disorders) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 11 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Flatulence (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 10 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 7
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 2
Nasopharyngitis (Infections and infestations) | 19 | 3
Pharyngitis (Infections and infestations) | 1 | 2
Rhinitis (Infections and infestations) | 6 | 2
Sinusitis (Infections and infestations) | 4 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 6
Urinary tract infection (Infections and infestations) | 12 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT03729362/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT03729362/SAP_001.pdf